CLINICAL TRIAL: NCT04935658
Title: Study of Analgesic Effect of Virtual Reality During Oocyte Retrieval in in Vitro Fecondation Protocols: Controlled Randomized Trial
Brief Title: Oocyte Retrieval and Virtual Reality (REVPO)
Acronym: REVPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOI 2020 VALDEYRON; 2020-A03233-36 (Other: ANSM)
Record Dates: First submitted 2021-05-25; First posted 2021-06-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Oocyte Retrieval; Pain; Fertilization in Vitro
Keywords: Reproductive Techniques, Assisted; Oocyte retrieval; Virtual reality; Medically Assisted Procreation; Pain; Analgesia
MeSH Terms: conditions — Pain; Helping Behavior; Agnosia | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: participants receive an intervention throughout the protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Group (Experimental): in this group, patients will use virtual reality during the oocyte retrieval plus the standard anesthesic procedure (local anesthesia)
  Interventions: Device: Hypnotic relaxation induced by virtual reality (device); Drug: local anesthesia
- Standard Group (Sham Comparator): in this group, patients will receive the standard anesthesic procedure during the oocyte retrieval wich is local anesthesia
  Interventions: Drug: local anesthesia

INTERVENTIONS:
Device: Hypnotic relaxation induced by virtual reality (device) — A virtual reality device will be install on the patient 3-5 minutes before the beginning of the oocyte retrieval. The device will be wearing by the patient during the entire intervention and 2 minutes after the end of the ponction.
  Arms: Virtual Reality Group
Drug: local anesthesia — standard anesthesic procedure

SUMMARY:
The aim of the study is to ass wether or not the use of virtual reality during oocyte retrieval provides a better pain relief for patients, compared to a standard analgesic procedure.

DETAILED DESCRIPTION:
Patients will be included during the consultation with the gynaecologist, whom will explain the protocol to the patient and give her the consent to sign.

The patient will be then randomized by a computer (using the software REDCAP) into either the experimental group or the standard group.

In the experimental group, a virtual reality device will be installed on the patient as soon as she arrives in the operating room, and the intervention will start after 3-5 minutes.

In both group, the patient will benefit of a local anesthesia in the vagina, and if they want it of an oral analgesic before the intervention.

Just at the end of the intervention, the pain will be evaluated orally by the nurse, using a Numeric Rating Scale. This consist of the Primary Outcome.

After the intervention, the gynaecologist will fill a form assessing his satisfaction concerning the use of virtual reality during the intervention (efficacy, security...) One hour after the intervention, the patient will fill a form about her self-estimation of the post-procedural pain and her satisfaction concerning the use of virtual reality.

The number of oocytes collected and the number of oocytes expected on the ultrasound monitoring will be gathered and a ratio will be calculated, in order to estimate the efficacy of the retrieval.

Five days after the intervention, the patient will have to fill a form evaluating her consumption of painkillers during the 48hours following the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 43 years
* First attempt of oocyte retrieval under local anesthesia in the context of a protocol for Medically Assisted Procreation

Exclusion Criteria:

* Former attempt of oocyte retrieval
* Poor oocyte stock : > 40 years AND low markers (AMH < 0.5-1.1 ng/ml OR AFC < 5-7)
* Unsteady epilepsia

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Pain during oocyte retrieval, assessed by NRS | day 0 (During the intervention for oocyte retrieval)
  Oral evaluation of pain during the intervention for oocyte retrieval, evaluated by a Numeric Rating Scale (NRS) : from 0 (meaning no pain at all) to 10 (meaning worse pain possible).

SECONDARY OUTCOMES:
Pain after oocyte retrieval, assessed by NRS | hour 1 (In the hour following the oocyte retrival)
  Written evaluation of pain after the intervention for oocyte retrieval, evaluated by a Numeric Rating Scale (NRS) : from 0 (meaning no pain at all) to 10 (meaning worse pain possible).
Painkillers consumption during the 48 hours following the oocyte retrieval. | Day 5
  Written auto-evaluation (questionnaire) of the amount and type of painkillers taken by the patient during the 48hours following the intervention
Patient satisfaction concerning the use of virtual reality during the oocyte retrieval | hour 1 (In the hour following the oocyte retrival)
  Written evaluation of the patient global satisfaction concerning the virtual reality during the oocyte retrieval. (2 questions : "Concerning the use of virtual reality during the oocyte retrieval, are you : very satisfied, little satisfied, not satisfied, not at all satisfied"; "if you had to re-take an oocyte retrieval, would you : do it again with virtual reality, do it again without virtual reality, do it under general anesthesia")
Gynaecologist satisfaction concerning the use of virtual reality during the oocyte retrieval | hour 1 (In the hour following the oocyte retrival)
  Written evaluation of the gynaecologist satisfaction concerning the use of virtual reality during the oocyte retrieval (4 questions : "Concerning the security during the oocyte retrieval, are you very satisfied, little satisfied, not satisfied, not at all satisfied", "Concerning the easiness of the oocyte retrieval, are you very satisfied, little satisfied, not satisfied, not at all satisfied", "During the oocyte retrieval, the patient seemed : very relaxed, relaxed, not relaxed, not at relaxed"; "as a whole, if this patient should re-take an oocyte retrieval, ould you recommend the use of virtual reality? Yes/No, can you tell us why in a few words")
Efficacy of the use of virtual reality during oocyte retrieval | hour 1 (In the hour following the oocyte retrival)
  Ratio between the number of oocytes collected during the retrieval compared to the number of oocytes expected on the ultrasound monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Camille Valdeyron, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No